CLINICAL TRIAL: NCT00961571
Title: A Single-Center, Phase II Trial of Sunitinib and Capecitabine in First Line Treatment of Patients With Metastatic Colorectal Cancer
Brief Title: Sunitinib and Capecitabine for First Line Colon Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unanticipated side effects and futility
Sponsor: Georgetown University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA61822D; 2008-308 (Other: IRB)
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; sunitinib; capecitabine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sunitinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sunitinib and cepecitabine (Experimental): Administration of sunitinib and capecitabine
  Interventions: Drug: sunitinib and capecitabine

INTERVENTIONS:
Drug: sunitinib and capecitabine — Sunitinib 37.5 mg po once daily Capecitabine 1000 mg po twice daily
  Other Names: Sunitinib, NSC 736511, Sutent; Capecitabine, Xeloda

SUMMARY:
This study is for patients with metastatic colorectal cancer who have not been treated with chemotherapy for their cancer. The purpose of this study is to find out if Capecitabine and Sunitinib can be used together to improve progression-free survival in colorectal cancer.

All patients will take two medicines (Sunitinib and Capecitabine) by mouth every day until their cancer gets worse.

DETAILED DESCRIPTION:
This is a single-center, open-label, one-arm study. Patients will be stratified by prior adjuvant therapy and ECOG performance status at study entry.

In this study, we propose to obtain PET scans at baseline, 2 weeks, 8 weeks and 24 weeks from the initiation of treatment. Response at 2 weeks, 8 weeks and 24 weeks will be correlated to progression-free survival, overall survival and response according to RECIST criteria.

We will collect plasma and urine samples from enrolled patients before and four weeks after sunitinib treatment. The samples will be analyzed and results correlated with patient clinical outcomes in order to explore the underlying mechanism of sunitinib induced hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, newly diagnosed metastatic colorectal cancer
* Measurable or evaluable disease in which surgical resection with curative intent is not possible
* No adjuvant chemotherapy within 6 months of enrollment
* No prior sunitinib or other receptor tyrosine kinase inhibitors
* 18 years of age or greater
* Anticipated survival of at least 6 months
* Ambulatory with an ECOG performance status of 0 or 1 and able to maintain weight
* Normal organ and marrow function
* Must agree to avoid pregnancy or fathering a child through out study participation
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Chemotherapy or radiotherapy within 6 months of enrollment
* Receiving any other investigational agents
* Known untreated brain metastases, uncontrolled seizure disorders, encephalitis, or multiple sclerosis
* Not able to ingest oral medications with normal absorption from the GI tract
* Uncontrolled hypertension
* History of severe/unstable angina, heart attack, congestive heart failure, transient ischemic attack, or stroke within 6 months of enrollment
* Cardiac dysrhythmias
* History of clinically significant bleeding within the past 6 months, including gross hemoptysis or hematuria, or underlying coagulopathy
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of study enrollment
* Current treatment with therapeutic doses of coumadin
* Concurrent malignancy other than colorectal cancer
* Known dihydropyrimidine dehydrogenase deficiency
* Uncontrolled intercurrent illness including ongoing or active infection or psychiatric illness that would limit compliance with study requirements.
* Pregnant and nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aiwu Ruth He, MD, Principal Investigator — Georgetown University
Locations (1):
- Lombardi Cancer Center at Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2007 to 2008, we treated patients with unresectable advanced colorectal cancer with Sunitnib 37.5 mg orally once daily and Capecitabine 1000 mg orally twice daily in a phase II clinical trial at Georgetown University Hospital
Period: Overall Study
Arm/Group | Sunitinib and Cepecitabine
Started | 50
Completed | 11 (high percentage of patient drop-off study prior cancer progression)
Not Completed | 39
Not completed — Physician Decision | 39

BASELINE CHARACTERISTICS:
Population: metastatic colon cancer who has not received 1st line systemic chemotherapy
Arm/Group | Sunitinib and Cepecitabine
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 67 [23 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) will be measured as the number of months between each patient's enrollment and his/her date of progression or date of death.
Time Frame: 36 months
Population: Progression-free survival (PFS) will be measured as the number of months between each patient's enrollment and his/her date of progression or date of death.
Measure: Median (Full Range); unit: months
Arm/Group | Sunitinib and Cepecitabine
Number analyzed (Participants) | 11
months | 18.35 [7.57 to 31.57]

ADVERSE EVENTS:
Arm/Group | Sunitinib and Cepecitabine
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 8/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib and Cepecitabine (N=11)
Hypoalbuminemia (Hepatobiliary disorders) | 5
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 1
Febrile neutropenia (General disorders) | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Nausea (General disorders) | 1
Neuropathy (Nervous system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3
GI Obstruction (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib and Cepecitabine (N=11)
Alkaline phosphatase (Gastrointestinal disorders) | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 2
Anorexia (Gastrointestinal disorders) | 4
AST, SGOT(serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 4
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1
Bruising (General disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dehydration (General disorders) | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dry Lips (General disorders) | 1
Dysphagia (difficulty swallowing) (General disorders) | 1
Edema: limb (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Hyperglycemia (Endocrine disorders) | 2
Hematoma (General disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 6
Hemorrhage, CNS (Blood and lymphatic system disorders) | 1
Hemorrhage, GI::Abdomen (Gastrointestinal disorders) | 1
Hemorrhage, GU::Urinary (Blood and lymphatic system disorders) | 1
Hemorrhage/Bleeding - Other (Blood and lymphatic system disorders) | 1
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 10
Lymphopenia (Blood and lymphatic system disorders) | 3
Hypermagnesemia (Blood and lymphatic system disorders) | 1
Mucositis/stomatitis (General disorders) | 2
Nausea (General disorders) | 5
Neurology - Other (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 3
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 7
Pain - Other (General disorders) | 2
Pain::Abdomen (General disorders) | 3
Pain::Back (General disorders) | 1
Pain::Urethra (Renal and urinary disorders) | 1
Platelets (Blood and lymphatic system disorders) | 4
Hypokalemia (Blood and lymphatic system disorders) | 1
Rash/desquamation (General disorders) | 1
Sweating (diaphoresis) (General disorders) | 1
Taste alteration (dysgeusia) (General disorders) | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Tremor (General disorders) | 1
Weight loss (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less